CLINICAL TRIAL: NCT03327363
Title: The Clinical Efficacy and Stability of Information and Communication Technology (ICT)- Based Centralized Monitoring System of Asthma Control Monitoring in Asthma Patients: a Prospective, Randomized Controlled, Multicenter Study
Brief Title: Information and Communication Technology (ICT)- Based Centralized Monitoring System of Asthma Control
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yeungnam University Hospital (Other)
Collaborators: Ministry of Trade, Industry & Energy, Republic of Korea (Other Government); Korea Evaluation Institute of Industrial Technology (Other); Daegu Metropolitan City, Korea (Other Government); ICT Clinical Trial Coordination Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ICT-RTM-P06 Asthma
Record Dates: First submitted 2017-05-30; First posted 2017-10-31 (Actual); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Asthma
Keywords: ICT based clinical trial,; eCRF; electronic -institutional review board (eIRB),; Centralized monitoring; contract research organization (CRO)
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: a prospective, randomized controlled, multicenter study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ICT base monitoring group (Experimental): In the ICT-based centralized monitoring group, both subjects and medical staff receive feedback regarding decreased lung function and exacerbation in asthma symptoms in the form of text messages
  Interventions: Device: Feedback using ICT based monitoring system
- control group (Placebo Comparator): Use standard asthma treatment
  Interventions: Device: Feedback using ICT based monitoring system

INTERVENTIONS:
Device: Feedback using ICT based monitoring system — In experimental group, the subjects the check their lung function using self FEV1 monitoring device (microlife PF-200). They send the information to central monitoring system(EDC systems). In case of decreased FEV1 compared with own average FEV1, the ICT based monitoring system send the feedback message to the subject and medical staffs.

SUMMARY:
The aims of this study is to evaluation of the clinical efficacy and stability of Information and Communication Technology (ICT)- based centralized monitoring system of asthma control monitoring in asthma patients. We planed to enroll 100 asthma patients (50 subjects using ICT systems, 50 controls). We will monitor the asthma control status, lung function, exacerbation rate and stability of ICT systems.

This study is based upon work supported by the Ministry of Trade, Industry & Energy (MOTIE, Korea) under industrial Technology Innovation Program (No. 10059066, 'Establishment of ICT Clinical Trial System and Foundation for Industrialization').

DETAILED DESCRIPTION:
This study has a multi- center, open- label, prospective and randomized clinical trial design. One hundred asthma patients who fill out the informed consent form are registered and randomized 1:1 into the ICT-based centralized clinical trial monitoring group (n=50) or the ambulatory follow-up group (n=50). The planned follow-up duration is 6 months. he ICT-based centralized clinical trial monitoring group is given home based spirometry and connecting system (gateway) equipped with personal identification system. Fingerprint registration is required in advance, so that it would be used for authentication before each use of spirometry. Symptom score and lung functions (FEV1, PEFR) obtained from gateway is saved, monitored, and sent out via a home-monitoring system. In the ICT-based centralized clinical trial monitoring group, feedback is sent to both patients and medical staff in the form of texts if there is a worsening of symptoms score and/or lung function.

Subjects are to make office visits after randomization at 4, (8), 12, (16, 20), and 24 weeks. (ICT group will not visit at the schedules in the brackets) Each visit requires measurement of Questionnaire (ACQ) lung functions.

ELIGIBILITY:
Inclusion Criteria:

* asthma patients diagnosed by doctors
* Current treatment with Inhaled corticosteroid or leukotriene receptor antagonist
* able to give written informed consent prior to participation in the study

Exclusion Criteria:

* Subjects with plan of administration or operation within study periods
* Unstable heart disease and psychical disorder
* refuse the monitoring

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-04-30 (Actual); Primary Completion 2018-11-30 (Estimated); Study Completion 2018-11-30 (Estimated)

PRIMARY OUTCOMES:
asthma control score | up to 24 weeks after enrollment
  Asthma control status will be checked using asthma control questionnaire (ACQ),
exacerbation rate | up to 24 weeks after enrollment
  exacerbation was defined as symptom score, and lung function
change of FEV1 | up to 24 weeks after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Hunn Jung Jin, MD, Study Chair — Yeungnam University Hospital
Locations (1):
- Yeungnam University Hospital, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No